CLINICAL TRIAL: NCT04776382
Title: Eye Movement Modeling Examples as a Teaching Tool for Epidural Block
Brief Title: Eye Movement Modeling Examples as a Teaching Tool
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: European e-Learning School in Obstetric Anesthesia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EESOA10
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Simulation Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Trainees of this group will watch an EMME (Eye Movement Modeling Examples) pre-recorded video, on where to focus their gaze while performing the epidural procedure in accordance with expert eye-tracking
  Interventions: Other: EMME (Eye Movement Modeling Examples)
- Control Group (No Intervention): Trainees of this group will not watch the pre-recorded video

INTERVENTIONS:
Other: EMME (Eye Movement Modeling Examples) — Trainees of this group will watch an EMME (Eye Movement Modeling Examples)-recorded video, on where to focus their gaze while performing the epidural procedure in accordance with expert eye-tracking
  Arms: Study Group

SUMMARY:
This study will evaluate whether eye-tracking assisted teaching (EMME, Eye Movement Modeling Examples) changes the visual patterns and improve the inexperienced trainee's performance in executing an epidural block on an epidural simulator.

DETAILED DESCRIPTION:
Eye Movement Modeling Examples (EMME) is the youngest topic within the field of applied eye-tracking research in Educational Science. These are video recordings of a model executing a task and explaining how he goes about that. On top of that, the model's eye movements are tracked and replayed on top of the video.

It addresses the question, how visual expertise could be trained with the help of instructional videos of real-world tasks that are explained by experts in the field. These videos include an overlay of these experts' visual focuses to support the learner in connecting the verbal explanation of the expert to the real-world complexity of the task. The aim of this study will be to evaluate whether eye-tracking assisted teaching may improve the novice, inexperienced, trainee's performance in executing an epidural block on an epidural simulator and may change its visual patterns as assessed by eye-tracking glasses.

The study will enroll 14 novice trainees who will be randomized into two equal groups to receive (study group) or to don't receive (control group) a pre-recorded video (intervention) containing the instructions on where to focus their gaze while performing the epidural procedure.

All the trainees (study and control group) will be asked to perform the epidural procedure using a standardized epidural simulator while wearing eye-tracking glasses.

For this study, the investigators will use a commercially available Tobii Pro Glasses 50 Hz wearable wireless eye tracker. This system can measure eye movements using cameras integrated into the eyeglasses which record the corneal reflection of infrared lighting to track pupil position, mapping the subject's focus of attention on video recordings of the subject's field of vision (gaze).

All the eye-tracked epidural procedures will be recorded immediately after accurate individual calibration, during which the participant, after wearing the glasses unit, focused on the center of the calibration target.

All the eye-tracking video-recordings will be stored and analyzed by using Tobii Pro Lab Software. The investigators will select six areas of interest (AOI), to define regions of a displayed stimulus, and to extract metrics specifically for those regions. The areas were the following: 1) point of the epidural needle at its insertion into the skin; 2) shaft of the epidural needle; 3) hub of the needle; 4) barrel of the syringe; 5) plunger of the syringe; 6) other fields of view.

ELIGIBILITY:
Inclusion Criteria:

* inexperienced trainees in anesthesia who have never performed an epidural block

Exclusion Criteria:

* trainees who have previously performed an epidural block

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-03-25 (Estimated); Primary Completion 2022-10-28 (Estimated); Study Completion 2022-10-28 (Estimated)

PRIMARY OUTCOMES:
Eye Fixations Numbers | up to 10 minutes
  Duration (seconds) of fixations for each area of interest and for each phase will be examined.
  Fixations are represented as discrete samples of almost stable points where the eye is looking. Their duration is the elapsed time between the start of the first fixation on the AOI until the end of the last fixation on the AOI. The duration of fixations for each area of interest and for each phase will be examined.
Eye Fixation duration | up to 10 minutes
  The number of fixations for each area of interest and for each phase will be examined.
  Fixations are represented as discrete samples of almost stable points where the eye is looking. The number of fixations for each area of interest and for each phase will be examined.

SECONDARY OUTCOMES:
Epidural attempt | up to 10 minutes
  An attempt will be defined as a complete withdrawal of the needle from the epidural simulator's skin and its reinsertion at the same or at a different interspace
Duration of the epidural procedure | up to 30 minutes
  The total duration of the procedure will be defined as the length of time between the insertion of the epidural needle into the skin of the simulator and the completion of the loss of resistance technique (finding of the epidural space).

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Capogna, MD, Study Director — European e-Learning School in Obstetric Anesthesia
Locations (1):
- EESOA srl, Roma, Italy

IPD SHARING:
Plan to Share IPD: No